CLINICAL TRIAL: NCT02681965
Title: A Randomized Controlled Trial, Using a Mail and Video-based Weight Loss Program for Overweight or Obese Stage I-IIIC Breast Cancer Survivors.
Brief Title: A Mail and Video-based Weight Loss Trial in Breast Cancer Survivors
Acronym: LEAN3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1410014716
Record Dates: First submitted 2016-02-10; First posted 2016-02-15 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer Survivorship; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LEAN (Experimental): Participants randomized to the weight loss program will initially receive the LEAN book, as well as a CD and flash drive with the LEAN videos (and internet link), a pedometer and the Log Book for recording their food intake and physical activity. Written instructions in the LEAN book will include recording daily diet and exercise in the logs. At the end of the study, participants will return, via a stamped addressed envelope, the logs to the study office so compliance can be assessed.
  Interventions: Behavioral: LEAN book/videos
- Waitlist Control (No Intervention): Participants randomized to the waitlist control study arm will be mailed the six-month questionnaires, which will include reporting of weight. On return of the 6-month questionnaires each woman will be provided with the entire weight loss program packet.

INTERVENTIONS:
Behavioral: LEAN book/videos — The intervention focuses on achieving long lasting lifestyle changes to achieve weight loss and maintenance. Women randomized to the weight loss program will receive the LEAN book, as well as a CD and flash drive with the LEAN videos (and internet link), a pedometer and the Log Book for recording their food intake and physical activity.
  Arms: LEAN

SUMMARY:
Proposed is a 6-month randomized controlled trial, in 200 overweight or obese Stage I-IIIC breast cancer survivors examining 6-month changes in: 1) body weight, 2) diet, 3) physical activity, and 4)quality of life in women randomized to receive the modified LEAN intervention compared to women randomized to wait-list control (i.e., the wait-list control will receive the modified LEAN intervention after completing the 6-month study).

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the effects of modifying the LEAN intervention (NCT02110641) to make it more cost effective by reducing or eliminating the counseling sessions. To guide the modification of the intervention one or more focus group sessions with former LEAN participants will be conducted. The purpose of these meetings will be to gain input on enhancing the LEAN book.

The LEAN book will be central to the modified intervention, but the LEAN book will be modified based on feedback from the focus group(s) and experience gained from the LEAN study. The reading level of the LEAN book will also be assessed to ensure acceptability to those with a low literacy level.

Once these changes have been finalized, the efficacy of the modified program will be tested using the methods described in the Brief Summary.

ELIGIBILITY:
Inclusion Criteria:

* Overweight individuals (BMI >= 25.0 kg/m2)
* Breast cancer survivors who have completed chemotherapy and/or radiation therapy
* Stage 0-III
* The ability to be physically able to exercise (e.g. walk at a moderate pace)
* Agree to random assignment to either group
* Give informed consent to participate in all study activities
* Accessible by telephone
* Able read and communicate in English

Exclusion Criteria:

* Pregnant or intending to become pregnant in the next year
* Recent (past 6 months) stroke or myocardial infarction
* Severe uncontrolled mental illness

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2016-03; Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Body weight (kg) | 6 Months
  A standard digital scale will be mailed to each participant along with the baseline packet to allow consistent measurement of weight by participants. Participants will weigh themselves. Body weight will be collected in kilograms (kg).

SECONDARY OUTCOMES:
Body weight (kg) | Baseline
  A standard digital scale will be used to measure participants at baseline. Body weight will be collected in kilograms (kg).
Body weight (kg) | 12 Months
  A standard digital scale will be mailed to each participant along with the baseline packet to allow consistent measurement of weight by participants. Participants will weigh themselves. Body weight will be collected in kilograms (kg).
Quality of Life (QOL) | Baseline
  QOL will be self-reported and collected at the baseline and 6-months. The Functional Assessment of Cancer Therapy-Breast (FACT-B) questionnaire will be administered to assess overall quality of life. The FACT-B measures physical, emotional, social, and functional well-being as well as quality of life issues specific to breast cancer survivors. The overall score will be used for assessment.
Quality of Life (QOL) | 6 months
  QOL will be self-reported and collected at the baseline and 6-months. The Functional Assessment of Cancer Therapy-Breast (FACT-B) questionnaire will be administered to assess overall quality of life. The FACT-B measures physical, emotional, social, and functional well-being as well as quality of life issues specific to breast cancer survivors. The overall score will be used for assessment.
Dietary Intake | Baseline
  The endpoint measures of diet change will be mean, group level changes in daily caloric intake, based on a 120-item food frequency questionnaire (FFQ) which was developed for the Women's Health Initiative Study and has been validated against 4-Day Food Records and 24-hour Dietary Recalls. The FFQ is used to generate the Healthy Eating Index score (HEI). The HEI will be used to assess dietary intake.
Dietary Intake | 6 months
  The endpoint measures of diet change will be mean, group level changes in daily caloric intake, based on a 120-item food frequency questionnaire (FFQ) which was developed for the Women's Health Initiative Study and has been validated against 4-Day Food Records and 24-hour Dietary Recalls. The FFQ is used to generate the Healthy Eating Index score (HEI). The HEI will be used to assess dietary intake.
Dietary Intake | 12 months
  The endpoint measures of diet change will be mean, group level changes in daily caloric intake, based on a 120-item food frequency questionnaire (FFQ) which was developed for the Women's Health Initiative Study and has been validated against 4-Day Food Records and 24-hour Dietary Recalls. The FFQ is used to generate the Healthy Eating Index score (HEI). The HEI will be used to assess dietary intake.
Physical Activity (Moderate) | Baseline
  Women will complete a physical activity questionnaire to assess their past six months of physical activity.10 Hours/week spent in different types (recreational, household, and occupation) and intensities (light, moderate, and vigorous-intensity) of activity will be computed over the past six months. Total minutes per week will be calculated from this survey for moderate and vigorous activity.
Physical Activity (Moderate) | 6 months
  Women will complete a physical activity questionnaire to assess their past six months of physical activity.10 Hours/week spent in different types (recreational, household, and occupation) and intensities (light, moderate, and vigorous-intensity) of activity will be computed over the past six months. Total minutes per week will be calculated from this survey for moderate and vigorous activity.
Physical Activity (Moderate) | 12 months
  Women will complete a physical activity questionnaire to assess their past six months of physical activity.10 Hours/week spent in different types (recreational, household, and occupation) and intensities (light, moderate, and vigorous-intensity) of activity will be computed over the past six months. Total minutes per week will be calculated from this survey for moderate and vigorous activity.
Physical Activity (Vigorous) | Baseline
  Women will complete a physical activity questionnaire to assess their past six months of physical activity.10 Hours/week spent in different types (recreational, household, and occupation) and intensities (light, moderate, and vigorous-intensity) of activity will be computed over the past six months. Total minutes per week will be calculated from this survey for moderate and vigorous activity.
Physical Activity (Vigorous) | 6 months
  Women will complete a physical activity questionnaire to assess their past six months of physical activity.10 Hours/week spent in different types (recreational, household, and occupation) and intensities (light, moderate, and vigorous-intensity) of activity will be computed over the past six months. Total minutes per week will be calculated from this survey for moderate and vigorous activity.
Physical Activity (Vigorous) | 12 months
  Women will complete a physical activity questionnaire to assess their past six months of physical activity.10 Hours/week spent in different types (recreational, household, and occupation) and intensities (light, moderate, and vigorous-intensity) of activity will be computed over the past six months. Total minutes per week will be calculated from this survey for moderate and vigorous activity.

CONTACTS AND LOCATIONS:
Overall Officials: Yale School of Medicine Irwin, Ph.D., Principal Investigator — MEPH Chronic Diseases, Yale School of Medicine
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided